CLINICAL TRIAL: NCT02593799
Title: Non-invasive Prediction of Esophageal Varices in Liver Cirrhosis: A Multicenter Observational Study
Status: Completed | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Dr., General Hospital of Shenyang Military Region
Other Study IDs: NIPEV-1
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Liver Cirrhosis; Esophageal and Gastric Varices
Keywords: Liver cirrhosis; Esophageal and Gastric Varices; Endoscopy
MeSH Terms: conditions — Liver Cirrhosis; Esophageal and Gastric Varices | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with esophageal varices: Esophageal varices were confirmed by endoscopy. They were divided into "any grade" and "high-risk" varices.
  Interventions: Procedure: Endoscopy
- Patients without esophageal varices: Patients without esophageal varices were divided into patients without "any grade" or "high-risk" varices.
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Upper gastrointestinal endoscopy to evaluate the presence of any grade varices and high-risk varices.

SUMMARY:
Esophageal variceal bleeding is one of the most lethal complications of liver cirrhosis. In the early stage of liver cirrhosis, the prediction of esophageal varices is very important for guiding the clinical decision making of primary prophylaxis of variceal bleeding.

DETAILED DESCRIPTION:
Esophageal variceal bleeding is one of the most lethal complications of liver cirrhosis. In the early stage of liver cirrhosis, the prediction of esophageal varices is very important for guiding the clinical decision making of primary prophylaxis of variceal bleeding. The investigators' recent systematic review evaluated the diagnostic accuracy of APRI, AAR, FIB-4, FI, King, Lok, Forns, and FibroIndex scores in predicting the presence of esophageal varices in liver cirrhosis. However, their diagnostic accuracy was low to moderate. Further study is warranted to establish a reliable score to predict the presence of high-risk esophageal varice in liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of liver cirrhosis.
2. Age and sex are not limited.
3. Etiology of liver cirrhosis is not limited.
4. Routine laboratory data.
5. Upper gastrointestinal endoscopy.

Exclusion Criteria:

1. Non-cirrhotic portal hypertension.
2. Malignancy.
3. Absent laboratory data.
4. A previous diagnosis of esophageal varices.
5. A previous history of variceal bleeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with liver cirrhosis who will firstly undergo the upper gastrointestinal endoscopy.
Sampling Method: Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation of biochemical data with esophageal varices in liver cirrhosis | 18 months
  The investigators firstly calculated the significant factors associated with the presence of esophageal varices, and then developed a score to predict the presence of esophageal varices in liver cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Guo, M.D., Principal Investigator — Department of Gastroenterology, General Hospital of Shenyang Military Area
Locations (17):
- China (17):
  - ANSTEEL Group Hospital, Anshan, Liaoning
  - Shuangshan Hospital of Anshan City, Anshan, Liaoning
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Friendship Hospital of Dalian City, Dalian, Liaoning
  - Central Hospital of Dandong City, Dandong, Liaoning
  - Central Hospital of Fushun City, Fushun, Liaoning
  - General Hospital of Mining Industry Group Fuxin, Fuxin, Liaoning
  - First Affiliated Hospital of Liaoning Medical University, Jinzhou, Liaoning
  - General Hospital of Liaoyang City, Liaoyang, Liaoning
  - Central Hospital of Panjin City, Panjing, Liaoning
  - General Hospital of Liaohe Oil Field, Panjing, Liaoning
  - Department of Gastroenterology, General Hospital of Shenyang Military Area, Shenyang, Liaoning
  - Central Hospital Affiliated to Shenyang Medical College, Shenyang, Liaoning
  - First Affiliated Hospital of Chinese Medical University, Shenyang, Liaoning
  - No. 1 of Department of Gastroenterology, Liaoning Provincial People's Hospital, Shenyang, Liaoning
  - No. 2 of Department of Gastroenterology, Liaoning Provincial People's Hospital, Shenyang, Liaoning
  - Shengjing Hospital of Chinese Medical University, Shenyang, Liaoning

REFERENCES:
- [Background] Deng H, Qi X, Guo X. Diagnostic Accuracy of APRI, AAR, FIB-4, FI, King, Lok, Forns, and FibroIndex Scores in Predicting the Presence of Esophageal Varices in Liver Cirrhosis: A Systematic Review and Meta-Analysis. Medicine (Baltimore). 2015 Oct;94(42):e1795. doi: 10.1097/MD.0000000000001795. PMID 26496312
- [Background] Qi X, Guo X, Li H, Liu X, Deng H. Knowledge about non-invasive diagnostic tests for varices in liver cirrhosis: A questionnaire survey to the Gastroenterology Branch of the Liaoning Medical Association, China. Gastroenterol Rep (Oxf). 2016 May;4(2):141-7. doi: 10.1093/gastro/gov031. Epub 2015 Jul 9. PMID 26159631
- [Derived] Qi X, Li Y, Wang R, Lin L, Li J, Wang L, Zheng S, Sun Y, Zhao L, Fu X, Wang M, Qiu X, Deng H, Hong C, Li Q, Li H, Guo X. Liaoning Score for Prediction of Esophageal Varices in Cirrhotic Patients Who Had Never Undergone Endoscopy: A Multicenter Cross-Sectional Study in Liaoning Province, China. Adv Ther. 2019 Aug;36(8):2167-2178. doi: 10.1007/s12325-019-00967-w. Epub 2019 May 15. PMID 31093864